CLINICAL TRIAL: NCT06840353
Title: The Effect of Intramuscular Ventrogluteal Injection Training Given by Pecha Kucha Method on Nursing Students' Knowledge, Skills and Satisfaction Levels: Randomized Controlled Trial
Brief Title: The Effect of Intramuscular Ventrogluteal Injection Training Given by Pecha Kucha Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Hilal Türkben Polat, Associate Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NEU-SKASBF-HTP-02
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Injection Site
Keywords: Pain; Nursing; Education; Injections, Intramuscular
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Single-blind parallel group randomized controlled trial
Who Masked: Investigator
Masking Description: The researcher will not know which group the participants were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Pecha Kucha training) (Experimental): Students will be given training on intramuscular injection for the Ventrogluteal region(VGR) using the Pecha Kucha training method. The 20-slide powerpoint presentation will last approximately 7 minutes. After the training, students will ; Complete the Knowledge Test for Intramuscular Injection to the VGR( 15 minutes after training). Students will complete the satisfaction scale after the training(15 minutes after training) . Afterwards, students will be taken to the Nursing Skills laboratory and will perform VG injection on a low-level intramuscular injection simulator(2 hour after training). The Skill Test for Intramuscular Injection to the VGR will be completed by an independent observer who is not a researcher while the student is performing the VG injection on simulator. Students' knowledge, skills and satisfaction will be measured again 30 days after the training with the same measurement tools.
  Interventions: Other: Experimental group (Pecha Kucha training)
- Control group (Standard Training Method) (No Intervention): Students assigned to the control group will be given intramuscular injection training for the Ventrogluteal region(VGR) with the Standard training method. The 30-slide powerpoint presentation will last approximately 20 minutes. After the training, students will ; Complete the Knowledge Test for Intramuscular Injection to the VGR( 15 minutes after training). Students will complete the satisfaction scale after the training(15 minutes after training) . Afterwards, students will be taken to the Nursing Skills laboratory and will perform VG injection on a low-level intramuscular injection simulator(2 hour after training). The Skill Test for Intramuscular Injection to the VGR will be completed by an independent observer who is not a researcher while the student is performing the VG injection on simulator. Students' knowledge, skills and satisfaction will be measured again 30 days after the training with the same measurement tools.

INTERVENTIONS:
Other: Experimental group (Pecha Kucha training) — Ventrogluteal injection training given to students using the Pecha Kucha training method
  Arms: Experimental group (Pecha Kucha training)

SUMMARY:
The aim of this study is to determine the effect of intramuscular Ventrogluteal injection training given with the Pecha Kucha method on the knowledge, skill and satisfaction levels of nursing students.

DETAILED DESCRIPTION:
Intramuscular injection is a very important intervention among basic nursing skills. Intramuscular injection technique to the ventrogluteal region is one of the safest injection techniques. In teaching this technique, both the knowledge and skills of the students can be increased by using different education methods. This research will be carried out to determine the effect of intramuscular ventrogluteal injection training given with the Pecha Kucha method on the knowledge, skill and satisfaction levels of nursing students.

Method: Data will be collected with the Introductory Information Form, Knowledge Test for Intramuscular Injection to the Ventrogluteal Region, Skill Test for Intramuscular Injection to the Ventrogluteal Region, Satisfaction Visual Analog (VAS) Scale. Data will be collected face to face between March 2025 and May 2025.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Fundamentals of Nursing course for the first time
* Being between the ages of 18-25
* Students who can speak and understand Turkish fluently.
* Students who accept to participate in the study voluntarily.

Exclusion Criteria:

* Students who have previously taken the Fundamentals of Nursing 1st year course.
* Students who are graduates of Health Vocational High School.
* Students who have transferred to the nursing department with the vertical transfer exam.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Knowledge Test for Intramuscular Injection to the Ventrogluteal Region | 15 minutes after training, 1 month after training
  It is a test with 24 propositions about VG injection. Propositions are answered as true, false and I have no idea. 1 point is given for each correct answer. The form was developed by the research team

SECONDARY OUTCOMES:
Skill Test for Intramuscular Injection to the Ventrogluteal Region | 2 hours later after training, 1 month after training
  It was prepared to measure the skill levels of students regarding VG injection application. It is a test that includes 33 application steps about VG injection and is evaluated out of 100 points in total. The student who performs each application step receives the score given in the test in return. The test is evaluated based on the total score. The form was developed by the research team
Satisfaction Visual Analog (VAS) Scale: | 15 minutes after training
  The scale consists of a horizontal or vertical line, scaled as 10 cm/100 mm. In this study, a form scored between 0-10 points in the horizontal feature will be used. In the satisfaction assessment, a score of 0 on the scale indicates no satisfaction, and a score of 10 indicates very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Türkben Polat, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No